CLINICAL TRIAL: NCT00485186
Title: Investigation of Gene Polymorphisms Influencing Steroid Synthesis and Action in Patients With Deficient Steroid Biosynthesis and Disorders of Sex Development
Brief Title: Gene Polymorphisms Influencing Steroid Synthesis and Action
Status: Withdrawn | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Felix Riepe, Prof. Dr., University Hospital Schleswig-Holstein
Other Study IDs: D429/05
Record Dates: First submitted 2007-06-08; First posted 2007-06-12 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Disorders of Sex Development; Congenital Adrenal Hyperplasia; Congenital Adrenal Hypoplasia; Adrenal Insufficiency; Mineralocorticoid Deficiency; Intersex
MeSH Terms: conditions — Disorders of Sex Development; Adrenal Hyperplasia, Congenital; Hypoadrenocorticism, Familial; Adrenal Insufficiency; Ovotesticular Disorders of Sex Development

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
The extend of steroid biosynthesis and action is mainly dependent on underlying genetic polymorphisms and gene mutations. These sequence variations in multiple genes involved in steroid biosynthesis and action cause different diseases (for example congenital adrenal hyperplasia or disorders of sex development). In addition, sequence variations in several other genes may influence the severity of a genetically caused disease of steroid biosynthesis or action. By this, the differences in an observed phenotype may be explained. Within the study all genes necessary for adrenal and gonadal steroid biosynthesis and several genes which are known to influence the action of steroid hormones will be analysed in patients with congenital disorders of adrenal and gonadal steroid biosynthesis, disorders of steroid action and disorders of sex development. The primary aim is to set up a correlation of the disease phenotype with the different genotypes detected.

ELIGIBILITY:
Inclusion Criteria:

* Disorders of Sex Development
* Congenital Adrenal Hyperplasia
* Congenital Adrenal Hypoplasia
* Adrenal Insufficiency
* Mineralocorticoid Deficiency
* Salt-loss

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion Criteria:
  * Disorders of Sex Development
  * Congenital Adrenal Hyperplasia
  * Congenital Adrenal Hypoplasia
  * Adrenal Insufficiency
  * Mineralocorticoid Deficiency
  * Salt-loss
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul-Martin Holterhus, MD, Study Chair — University Hospital Schleswig-Holstein; Felix G Riepe, MD, Principal Investigator — University Hospital Schleswig-Holstein